CLINICAL TRIAL: NCT04878575
Title: A Novel Multi-dimensional Prospective Study of the Gut-brain Axis Through Metabolic MRI, Metabolomics and Gut Microbiome to Discover Gene-microenvironment Interactions in Neurodevelopmental Disorders
Brief Title: A Multi-dimensional Prospective Study to Discover Gene-microenvironment Interactions in Neurodevelopmental Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201903105RINB
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Attention-Deficit Hyperactivity Disorder, Unspecified Type; Autism Spectrum Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — metabolite (blood) and intestinal microbial (stool)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD group: 120 ASD patients (aged 5-18 years)
  Interventions: Other: ASD diagnosis; Other: Psychiatric diagnosis
- ADHD group: 120 ADHD patients (aged 5-18 years)
  Interventions: Other: Psychiatric diagnosis
- TDC group: 120 age-, and sex-matched typically developing controls (TDC) will be recruited from the same geographic areas of the ASD/ADHD groups via referral by teachers or the invitation of participants without any psychiatric disorders
  Interventions: Other: Psychiatric diagnosis

INTERVENTIONS:
Other: ASD diagnosis — Autism Diagnostic Interview-revised (ADI-R) and Autism Diagnostic Observation Scale (ADOS)
  Groups: ASD group
Other: Psychiatric diagnosis — Kiddie Schedule for Affective Disorders & Schizophrenia (K-SADS) for DSM-5

SUMMARY:
This project is the first involving the two most common neurodevelopmental disorders, ASD and ADHD, as well as TDC to establish a multi-dimensional database (clinic, behavior, neurocognitive function, brain imaging, metabolomics, and microbiome) using the same methodology. Based on this integrated multi-dimensional databank, we anticipate exploring metabolic flows of the gut-brain axis during brain development and identifying the common and unique biomarkers of ASD and ADHD and high-risk materials related to their functions and the underlying mechanism. Moreover, distinguishing the characteristics of the gut microbiota, gastrointestinal disorders, and microbial flora dysbiosis also helps us, in turn, to accelerate the process of identifying biological treatments that can interfere or slow down the severity of cognitive impairments in neurodevelopmental disorders. Eventually, we anticipate finding the clinical and neurocognitive measures related to the direct or indirect influence of gut-brain signaling. Our findings are anticipated to improve the knowledge about neurodevelopmental disorders, enhance developing early detection, diagnosis, and treatment for ASD and ADHD, and contribute to precision medicine.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) and attention-deficit hyperactivity disorder (ADHD) are common neurodevelopmental disorders in Taiwan and worldwide (prevalence rate, ASD, 1%; ADHD, 3-10%), presenting as clinically and genetically heterogeneous disorders with early onset at childhood lasting to adulthood. Both disorders bring a tremendous impact on individuals, families, and society. Despite extensive studies on these two disorders, our knowledge about their pathogenetic mechanism is still minimal, and there are no biomarkers for effective prevention, early detection, diagnosis and biological treatment (ineffective in 30% ADHD patients, none for ASD). Although they have distinct symptom inclusion criteria and intervention, emerging evidence suggests that ASD and ADHD may share some genetic influences and susceptibility involving neuroanatomical phenotypes, cognitive deficits, and behavioral phenotypes. However, few studies have investigated these two disorders simultaneously. Moreover, the role of metabolomics and microbiome in neuropsychiatric disorders has drawn much attention recently. With the PI's long-term commitment to the neurocognitive/imaging/gene research ADHD and ASD in separate projects, our knowledge about these two disorders improved, but their underlying pathogenesis remains unclear. Hence, a multi-dimensional prospective gut-brain axis integration study highlighting the metabolism in the whole body to identify the common and unique factors of these two disorders and discover their gene-microenvironment interaction mechanism is extremely urgent and warranted.

Specific Aims:

1. To identify and compare the early environmental factors (e.g., maternal, and pre-, peri-, and post-natal factors) affecting the gut- microbiome, cognition, and brain structures and functions among the ASD, ADHD and TDC groups at ages of 4-12 years old;
2. To investigate the symptomatology, neuropsychology, neuroimaging, gut microbiome and metabolic biomarker signatures at Time 1 and Time 2 among the three groups while considering food, GI symptoms, and life style;
3. To investigate the changes (Time2-Time1), stability, and interactions of the symptomatology, neuropsychology, neuroimaging (MRI+MRS), gut microbiome and metabolic biomarker signatures in youths with ASD and ADHD as compared to TDC over a 2-4-year follow-up period.
4. To identify the predictors from the environmental (perinatal, food, lifestyle, family, school, neighborhood) and individual (behavior, gut microbiota, metabolomics, brain structure) factors for the neurocognitive/brain function and psychosocial outcomes in the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorder or attention-deficit hyperactivity disorder defined by the DSM-5 criteria, made by board-certificated child psychiatrists
* Ages range from 5 to 18
* Both parents are Han Chinese
* Subjects and their parents consented to have repeated assessments at 2 to 3 years later

Exclusion Criteria:

* Comorbidity with DSM-5 diagnoses of ADHD (TDC group), ASD (ADHD and TDC groups), schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorders, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use
* Comorbidity with neurological or systemic disorders
* Having a first degree relative who may have ASD based on family history method assessment (ADHD and TDC groups)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 120 ASD and 120 ADHD, aged 4-18 will be recruited from the Department of Psychiatry, National Taiwan Univeristy Hospital(NTUH), or the participants with ASD or ADHD from Taiwan's National Epidemiological Study of Child Mental Disorders (TNESCMD). 120 age-, and sex-matched typically developing controls (TDC) will be recruited from the same geographic areas of the ASD/ADHD groups via referral by teachers or the invitation of participants without any psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological functions: Continuous Performance Test(CPT) | 15 minutes
  The 4 dimensions of CPT: focused attention, hyperactivity/impulsivity, sustained attention, and vigilance
Neuropsychological functions: Cambridge Neuropsychological Test Automated Batteries(CANTAB) | 1.5 hours
  The 4 main cognitive components of CANTAB: Visual Memory, Attention, Working and Planning Memory (Executive Functions), and Decision Making
Structural neuroimaging: Diffusing spectrum imaging (DSI) | 1 hour
  DSI is performed using a pulsed-gradient spin-echo diffusion echo planar imaging (EPI) sequence with 102 diffusion-encoding directions
Multi-echo resting-state fMRI (rfMRI) | 1 hour
  rfMRI will be used to evaluate resting-state connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan